CLINICAL TRIAL: NCT04318379
Title: A Phase I Trial of an Immunotherapy (HCVax™) in Chronic Hepatitis C Infected Patients
Brief Title: Therapeutic Hepatitis C Virus Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GeneCure Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GC002
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Therapeutic HCV vaccine; HCV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose group (Experimental): Chronic HCV patients. Fifteen subjects will receive 1.0 ml of low dose vaccine at weeks 0, 8 and 16 through subcutaneous route.
  Interventions: Biological: HCVax
- High dose group (Experimental): Chronic HCV patients. Fifteen subjects will receive 1.0 ml of high dose vaccine at weeks 0, 8 and 16 through subcutaneous route.
  Interventions: Biological: HCVax

INTERVENTIONS:
Biological: HCVax — HCVax is a lentiviral vector encoding several HCV antigens

SUMMARY:
GC002 is a Phase I trial to evaluate the safety and the immune responses of a lentiviral based HCV immunotherapy (HCVax™) in chronic HCV patients.

DETAILED DESCRIPTION:
GC002 is a Phase I trial to evaluate the safety and the immune responses of a lentiviral based HCV immunotherapy (HCVax™) in chronic HCV patients. Chronic HCV patients will be enrolled sequentially into low dose and high dose groups. Following the vaccination subjects who received at least one vaccination will be followed up for safety and immunological response through week 28. All vaccine recipients will take part in a long-term safety follow-up for 6 months following the completion of the vaccine series to assess delayed adverse events.

Vaccination will first start at low dose. The investigators will enroll low dose group first. Two subjects will be staggering enrolled every 2 weeks. Following the assessment and review of prior vaccinations, if no vaccine definitely or probably-related severe adverse event (grade 3 or above) or SAE occurs the vaccination schedule for low dose and high dose will continue until complete enrollment.

Each subject will receive HCVax™ vaccine at 0, 8, 16 weeks through subcutaneous route. Following vaccination subjects will have clinical, immunological and virologic assessments throughout the 28-week study.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of chronic hepatitis C infection based on serum positivity for HCV RNA for at least 6 months interval. HCV genotype will be recorded. All genotypes will be eligible.
2. Patients who are not under DAA treatment.
3. Liver fibrosis (by Metavir stage F1 or F0) within one year of the screening visit, documenting extent of liver disease consistent with chronic hepatitis C with evidence of inflammation and/or fibrosis. Fibrosis scaling is based on an ultrasound based elastography (FibroScan, Echosen, Paris France) with cutoff of 7.5 kPa or liver biopsy.
4. Screening laboratory values within institutional normal range, with the exception of liver enzymes ≤ 3 ULN and bilirubin <1.5 ULN, or judged to be not clinically significant by clinical investigator.
5. Ability and willingness of subject to give written informed consent.
6. Negative pregnancy test on the day prior to each vaccination.
7. Willingness to use adequate contraception by study participants. Subjects must agree not to participate in a conception process (e.g., active attempts to become pregnant or to impregnate, sperm donation, or in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, subjects must use a form of contraception as listed below while on study vaccine and for 60 days after stopping study vaccine. Women without reproductive potential (i.e., have reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation) or women whose male partner has undergone successful vasectomy with documented azoospermia or has documented azoospermia for any other reason, are eligible without requiring the use of contraception.

Exclusion Criteria:

1. History of decompensated liver disease, including but not restricted to, portal hypertension as manifested by a known history of gastroesophageal varices, variceal bleeding, ascites or encephalopathy, histopathologic or clinical evidence of cirrhosis, hepatocellular carcinoma, or renal impairment consistent with hepatorenal syndrome; history of significant other non-HCV chronic liver disease, i.e. alcoholic hepatitis, autoimmune hepatitis.
2. History of hematologic disease (e.g., cryoglobulinemia, lymphoma), renal disease, dermatologic disease (e.g., lichen planus, porphyria cutanea tarda).
3. Seropositive for hepatitis B surface antigen (HBsAg) or HIV-1 antibody.
4. Autoimmune diseases or clinically serious cardiac, pulmonary, gastrointestinal, hepatic, renal or neurologic disease, which in the opinion of the investigator will compromise ability to participate in the study.
5. Previous receipt of any HCV experimental vaccine.
6. Pregnancy and breast-feeding.
7. Prior or current systemic cancer chemotherapy.
8. Investigational agents and immunomodulators (cyclosporine, hematological growth factors, systemic corticosteroids, interleukins or interferons) within 90 days prior to study entry. NOTE: Subjects may not be on antiretroviral agents not yet approved by the FDA as part of a clinical trial or expanded access program.
9. Anaphylaxis or allergy to vaccine components.
10. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
11. Any other serious diseases other than HCV infection including current or recent (within 5 years) cancers.
12. Liver fibrosis with Metavir stage F2 or above.
13. Subjects with diabetes mellitus, who are at higher risk for more rapid progression of fibrosis.
14. Subjects who are immunocompromised or immunosuppressed due to disease or medications.
15. Subjects with any laboratory abnormalities Grade 3 or greater.
16. Women who are lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of a therapeutic HCV vaccine in chronic HCV patients | 40 weeks
  Frequency and severity of adverse events, laboratory abnormalities, local and systemic reactogenicity signs and symptoms following vaccinations.

SECONDARY OUTCOMES:
To evaluate the immunogenicity of a therapeutic HCV vaccine in chronic HCV patients | 40 weeks
  Magnitude of IFN-γ & IL-2 producing CD4+ and CD8+ T cells to HCV core peptides pools at weeks 8, 16, and 24.
Virologic response | 40 weeks
  Sustained viral response (SVR) will be defined as negative HCV RNA result using an assay that has sensitivity of 25 IU or less per milliliter at 12 weeks after the end of vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Final data will be published

REFERENCES:
- [Background] Tung FY, Tung JK, Pallikkuth S, Pahwa S, Fischl MA. A therapeutic HIV-1 vaccine enhances anti-HIV-1 immune responses in patients under highly active antiretroviral therapy. Vaccine. 2016 Apr 27;34(19):2225-32. doi: 10.1016/j.vaccine.2016.03.021. Epub 2016 Mar 19. PMID 27002500